CLINICAL TRIAL: NCT01382641
Title: Relevance of Eye Dominance in the Selection of Patients Suitable for Treatment With Monovision After Cataract Surgery
Brief Title: Show Improved Vision With the HOYA AF-1 Aspheric Intraocular Lens After Cataract Surgery
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Innovative Medical (Industry)
Responsible Party: James McDonald, McDonald Eye Associates, PA
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Hoya AF-1
Record Dates: First submitted 2011-06-03; First posted 2011-06-27 (Estimated); Last update posted 2011-10-06 (Estimated); Status verified 2011-10

CONDITIONS: Cataracts
Keywords: Cataract surgery
MeSH Terms: conditions — Cataract

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Hoya AF-1 IOL (Other)
  Interventions: Device: Hoya AF-1 IOL
- Revital Vision (Other)
  Interventions: Device: Revital vision

INTERVENTIONS:
Device: Hoya AF-1 IOL — The patients will be assessed for three months
  Arms: Hoya AF-1 IOL
Device: Revital vision — The patients will be assessed for three months.
  Arms: Revital Vision

SUMMARY:
The doctors participating in this study are looking to show improved vision with the HOYA AF-1 aspheric intraocular lens after cataract surgery. They will also study the use of Revital Vision (neuro-sensory testing) in providing the highest potential for improved vision.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must desire to pursue some type of mono-vision fit, mono-vision lasik, or mono-vision cataract surgery with lens implant.
2. Patients must be candidates for intraocular lens implantation for the correction of aphakia following extracapsular cataract extraction by phaco-emulsification.
3. Patients must be candidates for bilateral implantation and desiring post-operative spectacle independence through targeted mono-vision.
4. Patients must have less than 1.50 diopters of corneal astigmatism
5. Patients must have the potential for best corrected visual acuity of 20/30 or better in each eye.
6. Patients must have the mental capacity to cooperate when undergoing a detailed postoperative refractive examination.
7. Patients must be an adult.
8. Patients must provide written informed consent for cataract surgery.
9. Patients must be willing and able to return for scheduled follow-up examinations for a period of 3 months (post-second eye) post-operatively.
10. Patients must be willing and able to provide feedback to various survey questions regarding overall satisfaction and ease of adaptation to mono-vision and range of vision, etc.

Exclusion Criteria:

1. Patients with 1.50 diopters or more of corneal astigmatism
2. Patients requiring a lens power less than 6 D or greater than 30 D
3. Patients with any anterior segment pathology (chronic uveitis, iritis, iridocyclitis, rubeosis iridis, corneal dystrophy or corneal degeneration, tear film deficiency, poor pupil dilation, etc.).
4. Patients with uncontrolled glaucoma or who require current treatment for glaucoma, or with visual field loss as a result of glaucoma.
5. Patients with retinal pathology or a history of retinal detachment.
6. Patients with proliferative diabetic retinopathy, macular degeneration, or other degenerative visual disorders.
7. Patients with a history of previous ocular surgery including corneal refractive surgery.
8. Patients with congenital bilateral cataracts.
9. Patients with marked microphthalmos or aniridia.
10. Patients who have only one functioning eye.
11. Patients who do not have the potential for visual acuity of 20/30 or better in each eye.
12. Patients lacking intact binocular vision.
13. Patients who do not have an intact capsulorhexis and posterior capsular bag at the time of cataract removal and lens implantation.
14. Patients who have incomplete or damaged zonules, or who have zonular rupture during cataract removal.
15. Patients with pupils greater than 7mm

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2010-09; Primary Completion 2011-12 (Estimated); Study Completion 2011-12 (Estimated)

PRIMARY OUTCOMES:
Measuring Ocular Dominance | 3 months
Overall post surgical outcomes | 3 months

SECONDARY OUTCOMES:
Measuring visual acuities | 3 months

CONTACTS AND LOCATIONS:
Locations (1):
- McDonald Eye Associates, PA, Fayetteville, Arkansas, United States